CLINICAL TRIAL: NCT00783731
Title: Low Dose of Midazolam is Superior to Conventional Dose for Rapid Sequence Intubation in Emergency Department (ED)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Purpose: Treatment
Other Study IDs: RSI study
Record Dates: First submitted 2008-10-30; First posted 2008-11-03 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Intubation
Keywords: intubation
MeSH Terms: interventions — Midazolam

ARMS (1):
- Low dose midazolam (Experimental)
  Interventions: Drug: Low dose midazolam

INTERVENTIONS:
Drug: Low dose midazolam

SUMMARY:
Midazolam has been used in rapid sequence intubation for a long time, and the recommended dose is 0.1mg/kg. In some studies, however, the reduced dose has been used with the concern of hemodynamic instability. We would like to investigate that the low dose midazolam could be used rather than the standard recommended dose, and also compare it to the etomidate, recently used sedatives, with respect to the side effects and the easy performance of intubation.

ELIGIBILITY:
Inclusion Criteria:

* patients who need rapid sequence intubation in emergency room

Exclusion Criteria:

* in hypotension(systolic blood pressure less than 90 mmHg
* severe trauma patients
* pregnant
* allergic to midazolam, etomidate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2008-10; Primary Completion 2010-10 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Emergency room, Seongnam-si, Gyeonggi-do
  - Boramae Medical Center, Seoul